CLINICAL TRIAL: NCT06698003
Title: A Phase 2 Study for Screening and Prevention of Adult T-cell Leukemia/Lymphoma With Mogamulizumab in High-Risk Carriers of HTLV-1
Brief Title: A Study of Mogamulizumab to Prevent Adult T-cell Leukemia/Lymphoma in People With HTLV-1
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 21-486
Record Dates: First submitted 2024-11-18; First posted 2024-11-20 (Actual); Last update posted 2025-03-04 (Actual); Status verified 2025-03

CONDITIONS: T-Cell Leukemia/Lymphoma, Adult; T-cell Leukemia/Lymphoma; T-cell Leukemia; Lymphoma
Keywords: T-Cell Leukemia/Lymphoma, Adult; T-cell Leukemia/Lymphoma; T-cell leukemia; Lymphoma; Mogamulizumab; HTLV-1; Memorial Sloan Kettering Cancer Center; 21-486
MeSH Terms: conditions — Precursor T-Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, T-Cell; Lymphoma | interventions — mogamulizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cohort 1 (Experimental): Cohort 1: 0.3 mg/kg of mogamulizumab every 12 weeks, for 2 total doses
  Interventions: Drug: Mogamulizumab
- Cohort 2 (Experimental): Cohort 2: 0.3 mg/kg of mogamulizumab every 6 weeks, for 4 total doses
  Interventions: Drug: Mogamulizumab

INTERVENTIONS:
Drug: Mogamulizumab — Cohort 1: 0.3 mg/kg of mogamulizumab every 12 weeks, for 2 total doses Cohort 2: 0.3 mg/kg of mogamulizumab every 6 weeks, for 4 total doses

SUMMARY:
The purpose of this study is to find out whether the study drug mogamulizumab is effective in preventing the development of adult T-cell leukemia/lymphoma (ATL) in people who are at higher risk for this type of cancer because they are infected with the HTLV-1 virus and because of changes seen in some of their immune system cells called T-cells.

ELIGIBILITY:
Inclusion Criteria:

Screening Cohort (US patients only):

* Age ≥18 years when informed consent is obtained
* Has freely given written informed consent to participate in the study

Treatment Cohorts (Cohorts 1 and 2):

* Positive for anti-HTLV-1 antibody in the serum using an FDA approved assay for US patients (Avioq HTLV-I/II Microelisa System). UK patients should use UK Accreditation Service (UKAS) accredited tests, Abbot Architect ELISA Serology Screening assay and confirmatory serology Western Blot (performed at Public Health England, Virus Ref Dept, Colindale).
* High-risk phenotype (PVL≥8% of PBMC)
* Age ≥18 years when informed consent is obtained
* Primary organ functions are stable

  * Neutrophil count: ≥ 1000/mm3, unless patient has diagnosis of ethnic neutropenia
  * Platelets: ≥100,000/mm3
  * Hemoglobin: ≥9.0 g/dL
  * Serum aspartate aminotransferase (AST): ≤1.5x upper limit of normal (ULN)
  * Alanine aminotransferase (ALT): ≤1.5x ULN
  * Total bilirubin: ≤1.5x ULN
  * Serum creatinine (Cr): ≤1.5x ULN
  * Blood oxygen saturation (SpO2): ≥90%
* Electrocardiogram (ECG): No abnormal findings requiring treatment are observed
* Has freely given written informed consent to participate in the study
* For females of reproductive potential: use of effective contraception during treatment and for at least 3 months after completion of mogamulizumab therapy. For males who have sexual intercourse with females of reproductive potential: use of effective contraception during treatment and for at least 3 months after completion of mogamulizumab therapy.

Exclusion Criteria:

In order to protect subjects and avoid any problems in evaluating the study drug, patients who meet any of the following criteria should be excluded from enrollment in the study, in either screening or treatment cohorts:

* Patients with a history of any of the following:

  * Neutrophil count: ≤1000/mm3, unless patient has diagnosis of ethnic neutropenia
  * Acute or chronic hepatitis or hepatic cirrhosis, other than patients with positive antibodies and negative PCR as noted in criteria #11 and #12 below.
  * Tuberculosis or with active tuberculosis
  * Myocardial infarction within 12 months prior to the date of enrollment
  * Allergic reaction to administration of antibody drug products
  * Other cancers. Patients with a history of a localized solid tumor who received definitive, curative treatment and who have been without evidence of disease for 5 years prior to enrollment will be able to enroll in the study. Patients with radically resected basal cell carcinoma of the skin, squamous cell carcinoma (except malignant melanoma), noninvasive cervix carcinoma, carcinoma in situ in the gastrointestinal tract or corpus of the uterus, localized thyroid cancer, and localized renal cell carcinoma will be able to enroll in the study if they are determined to be completely cured, even if within 5 years of enrollment.
* Prior treatment with immunosuppressants or interferon alpha products within 6 months prior to the date of enrollment
* Serious complications (heart failure, lung disease, renal failure, hepatic failure, uncontrolled diabetes mellitus, etc.)
* History of an active autoimmune disease that has required systemic treatment in past 2 years (ie, with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (eg, thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency) is not considered a form of systemic treatment and is allowed.
* Any ailment that could be exacerbated by the administration of KW-0761, in the judgment of the Principal Investigator or co-Investigator
* Diagnosis of ATL
* Women who are pregnant, breastfeeding, who may be pregnant, or wish to bear children while receiving treatment or within 3 months of last dose of mogamulizumab
* Patients who have taken multivitamins (Alinamin, vitamin C, etc.) or supplements such as fucoidan, catechin, and pentosan polysulfate within 2 weeks prior to the date of enrollment
* Prior treatment with other study drugs within 4 months prior to giving informed consent
* Complications of spinal cord compressive lesions such as cervical spine disease, disc herniation, and ossification of the yellow ligament
* Uncontrolled psychiatric disorder, epilepsy, or dementia
* Positive test for Hepatitis B surface antigen or HBV-DNA (using real-time PCR). Positive Hepatitis B core antibody is permitted if HBV-DNA PCR is negative and the patient remains on prophylaxis during study.
* Positive test for Hepatitis C virus antibody, unless Hepatitis C PCR is negative.
* Positive test for HIV antibody, unless undetectable HIV RNA > 6 months and CD4 within normal limits per institutional standard.
* Patients considered unqualified to participate in the study by the Principal Investigator or co-Investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 134 (Estimated)
Dates: Start 2024-11-15 (Actual); Primary Completion 2029-11-15 (Estimated); Study Completion 2029-11-15 (Estimated)

PRIMARY OUTCOMES:
Minimum dose and schedule of mogamulizumab to reduce the proviral load by ≥75% | 6 months from baseline
  To define the minimum efficacious dose and schedule of mogamulizumab to reduce the proviral load by ≥75% by pre-emptive treatment of HTLV-1 carriers with a limited course of mogamulizumab. The minimum efficacious dose will maintain ≥75% reduction in PVL from baseline levels for a minimum 6 months post completion of preemptive treatment with a limited course of mogamulizumab.

CONTACTS AND LOCATIONS:
Overall Officials: Steven Horwitz, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (7):
- United States (7):
  - Memorial Sloan Kettering at Basking Ridge (All protocol activities), Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth (All protocol activities), Middletown, New Jersey
  - Memorial Sloan Kettering Bergen (All Protocol Activities), Montvale, New Jersey
  - Memorial Sloan Kettering Cancer Center @ Suffolk-Commack (All protocol activities), Commack, New York
  - Memorial Sloan Kettering Westchester (All protocol activities), Harrison, New York
  - Memorial Sloan Kettering Cancer Center (All Protocol Activities), New York, New York
  - Memorial Sloan Kettering Nassau (All protocol activities), Uniondale, New York

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org